CLINICAL TRIAL: NCT03808662
Title: Precision Radiation for OligoMetastatIc and MetaStatic DiseasE (PROMISE)-004: Consolidative Use of Radiotherapy to Block (CURB) Oligoprogression
Brief Title: Randomized Study of Stereotactic Body Radiation Therapy (SBRT) in Patients With Oligoprogressive Metastatic Cancers of the Breast and Lung
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-431
Record Dates: First submitted 2019-01-16; First posted 2019-01-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: TNBC - Triple-Negative Breast Cancer; Triple Negative Breast Cancer; NSCLC; NSCLC Stage IV; Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Metastatic; NSCLC Stage IV Without EGFR/ALK Mutation
Keywords: SBRT; Stereotactic Body Radiotherapy; Non-hematology metatstatic cancer; non-CNS oligo-progressive disease; intracranial metastatic disease; Memorial Sloan Kettering Cancer Center; 18-431
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Early Stereotactic Body Radiotherapy/SBRT (Experimental): SBRT to all oligoprogressive sites
  Interventions: Radiation: Sterotactic Body Radiotherapy/SBRT
- Arm 2:Standard of Care (Active Comparator)
  Interventions: Drug: Standard of care

INTERVENTIONS:
Radiation: Sterotactic Body Radiotherapy/SBRT — In general, it is recommended using 9-10 Gy x 3 or 10 Gy x 5 fractions given every other day. Physicians should try to give the highest BED whenever possible while respecting normal tissue tolerance. All lesions are recommended to receive a biologically effective dose (BED) of 60 Gy or higher (BED10≥70), assuming α/β ratio of 10 and using the linear-quadratic model: BED = nd x [1 + d/(α/β)] where n is number of fractions and d is dose per fraction. Sometimes BED ≥80 Gy is preferred, with lower doses ≥50 Gy allowed at the discretion of the treating physician for concerns about normal tissue toxicity.
  Arms: Arm 1: Early Stereotactic Body Radiotherapy/SBRT
Drug: Standard of care — Standard of care per physician discretion
  Arms: Arm 2:Standard of Care

SUMMARY:
The purpose of this study is determine if receiving stereotactic body radiation(SBRT) when participants' metastatic tumors have just begun to grow increase the length of time before disease gets worse

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing and able to provide informed consent
* Metastatic disease detected on imaging and histologically confirmed:

Triple negative breast cancer TNBC (ER <1%, PR <1%, her-2-neu 0- 1+ by IHC or FISH-negative or as determined by MD discretion)

OR NSCLC (without known EGFR mutation or ALK/ROS1 rearrangement)

OR Other high-risk breast cancer (per physician's discretion) progressed on hormone or systemic therapy, regardless of ER/HER2 status

OR NSCLC with EGFR, ALK, or ROS1 targetable molecular alterations with disease progression on first-line tyrosine kinase inhibitor

Note:

* Biopsy of metastasis prior to enrollment is per treating physician's discretion per standard of care. It is preferred but not required.
* These patients are selected for the study given the similar survival outcomes when given standard of care therapies
* Patient has received at least first-line prior treatment with systemic therapy (either cytotoxic or targeted, including maintenance therapies).
* Patients who received prior immunotherapy are allowed.
* Patients who had any prior radiation therapy near or overlapping with the oligoprogressive sites are allowed to enroll.
* Patients with the following medical conditions precluding them from participating in other systemic therapy or drug trials are allowed:
* active liver disease, including viral or other hepatitis, or cirrhosis
* any other significant medical condition not under control, including any acute coronary syndrome within the past 6 months.
* a permanent pacemaker
* a QTc > 480 ms in the baseline EKG
* peripheral neuropathy of grade >/= 2 per NCI CTCAE
* history or known autoimmune disease
* current chronic systemic steroid therapy or any immunosuppressive therapy
* history of primary immunodeficiency or solid organ transplant
* known positive human immunodeficiency virus (HIV), chronic or active hepatitis B or C, or active hepatitis A
* active infection requiring systemic antibiotic therapy
* Patients can have more than 5 metastases but can only have 1-5 oligo-progressive lesions.
* Oligoprogression, defined as Response Evaluation Criteria in Solid Tumors (RECIST) or Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) documented progression in up to 5 individual lesions

Using Response Evaluation Criteria in Solid Tumors (RECIST) Criteria as a guide:

1. At least a 20% increase in the sum of the longest diameter (LD) of the lesion, taking as reference the smallest sum LD recorded since the last imaging OR
2. The appearance of one or more new lesions OR
3. New/malignant FDG uptake in the absence of other indications of progressive disease or an anatomically stable lesion OR
4. >/= 5mm increase in the diameter sum of the lesion

OR

Using Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) as a guide:

1. >30% increase in 18F-FDG SUV peak, with >0.8 SUV units increase in tumor SUV from the baseline scan in pattern typical of tumor and not of infection/treatment effect OR
2. Visible increase in the extent of 18F-FDG tumor uptake OR
3. New 18F-FDG avid lesions typical of cancer (including new bone lesion) and not related to treatment effect and/or infection

OR

Development of a new soft tissue metastatic lesion at least 5mm in size or any new bone metastasis

OR

Progressive enlargement of a known metastasis on 2 consecutive imaging studies at least 2 months apart with a minimum 5mm increase in size

* All sites of oligoprogression can be safely treated
* Maximum 5 progressing metastases in any single extra-cranial organ system (i.e. lung, liver, bone)

  a. If the clinical scenario deem that other forms of local therapy may be more suitable for the metastatic disease, such as surgical resection and interventional radiology-guided ablation, patients would be able to undergo other forms of local therapy with discussion with the PI
* No restriction on the total number of metastases
* Note: If the clinical scenario deem that other forms of local therapy may be more suitable for the metastatic disease, such as surgical resection and interventional radiology-guided ablation, patients would be able to undergo other forms of local therapy with discussion with the PI.
* For patients with brain metastases and oligoprogression elsewhere where stereotactic radiation to the brain is warranted, the brain lesions can be treated prior to randomization. This will not be counted toward the 5 progressive lesions.
* Any symptomatic metastatic sites requiring prompt palliative radiation (e.g. cord compression) can also be treated with standard of care radiation prior to randomization. This will not be counted toward the 5 progressive lesions.

  1. If the clinical scenario deem that other forms of local therapy may be more suitable for the metastatic disease, such as surgical resection and interventional radiology-guided ablation, patients would be able to undergo other forms of local therapy with discussion with the PI.

Exclusion Criteria:

* Pregnancy.
* Leptomeningeal disease.
* Serious medical comorbidities precluding radiotherapy, such as ataxia-telangiectasia or scleroderma.
* Any other condition which in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 52 weeks after final participant is enrolled
  To study if the addition of early SBRT to extra-cranial oligo-progressive metastatic disease could prolong PFS compared to no SBRT. PFS is defined as the time from randomization to disease progression or death.

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Riaz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (9):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Fred Hutchinson Cancer Research Center (Data Analysis Only), Seattle, Washington
- Princess Margaret Hospital/Ontario Cancer Institute (Data Analysis Only), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Tsai CJ, Yang JT, Shaverdian N, Patel J, Shepherd AF, Eng J, Guttmann D, Yeh R, Gelblum DY, Namakydoust A, Preeshagul I, Modi S, Seidman A, Traina T, Drullinsky P, Flynn J, Zhang Z, Rimner A, Gillespie EF, Gomez DR, Lee NY, Berger M, Robson ME, Reis-Filho JS, Riaz N, Rudin CM, Powell SN; CURB Study Group. Standard-of-care systemic therapy with or without stereotactic body radiotherapy in patients with oligoprogressive breast cancer or non-small-cell lung cancer (Consolidative Use of Radiotherapy to Block [CURB] oligoprogression): an open-label, randomised, controlled, phase 2 study. Lancet. 2024 Jan 13;403(10422):171-182. doi: 10.1016/S0140-6736(23)01857-3. Epub 2023 Dec 14. PMID 38104577
- [Derived] Lee J, Koom WS, Byun HK, Yang G, Kim MS, Park EJ, Ahn JB, Beom SH, Kim HS, Shin SJ, Kim K, Chang JS. Metastasis-Directed Radiotherapy for Oligoprogressive or Oligopersistent Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2022 Jun;21(2):e78-e86. doi: 10.1016/j.clcc.2021.10.009. Epub 2021 Nov 18. PMID 34903471
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org